CLINICAL TRIAL: NCT03287388
Title: MRI Measurement of the Effects of Moderate Versus Deep Neuromuscular Blockade on the Abdominal Working Space During Laparoscopic Surgery in a Prospective Cohort Study.
Brief Title: MRI Measurement of the Effects of Deep Neuromuscular Blockade on the Abdominal Working Space During Laparoscopy
Acronym: RELAX-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63227.091.17
Record Dates: First submitted 2017-09-04; First posted 2017-09-19 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Block; Surgery
Keywords: Laparoscopic surgery; Abdominal working space; Moderate neuromuscular blockade; Deep neuromuscular blockade; MRI measurement
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: Each patient wil serve as its own control:
  Each patient will start without neuromuscular blockade (phase 1), followed by moderate neuromuscular blockade (phase 2) and deep neuromuscular blockade (phase 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Rocuronium (Experimental): Phase 1: no neuromuscular blockade
  Interventions: Procedure: No Rocuronium
- Rocuronium (moderate NMB) (Experimental): Phase 2: moderate neuromuscular blockade (TOF 1-3)
  Interventions: Drug: Rocuronium (moderate NMB)
- Rocuronium (deep NMB) (Experimental): Phase 3: deep neuromuscular blockade (PTC 0-1)
  Interventions: Drug: Rocuronium (deep NMB)

INTERVENTIONS:
Procedure: No Rocuronium — Phase 1: The patient will undergo a routine MRI-abdomen without neuromuscular blockade: TOF ratio =1.
  Other Names: No neuromuscular blockade
  Arms: No Rocuronium
Drug: Rocuronium (moderate NMB) — Phase 2: Rocuronium will be titrated to a moderate NMB (TOF 1-3), monitored by TOF-watch. When an adequate moderate NMB is achieved, the patient will undergo a second MRI-abdomen.
  Other Names: Moderate neuromuscular blockade (Rocuronium)
  Arms: Rocuronium (moderate NMB)
Drug: Rocuronium (deep NMB) — Phase 3: The patient receives a bolus of 1.2 mg/kg rocuronium (adjusted to ideal body weight), to assure a deep or intense NMB (PTC 0-1). Then the patient will undergo the final, third MRI scan of the abdomen.
  Other Names: Deep neuromuscular blockade (Rocuronium)
  Arms: Rocuronium (deep NMB)

SUMMARY:
During laparoscopy, a surgical working space is obtained by creation of a pneumoperitoneum. Optimal surgical conditions are essential to ensure the patient's safety. A meta-analysis on studies comparing the influence of deep and moderate neuromuscular blockade (NMB) on the quality of the surgical space conditions during laparoscopy (1), showed that compared to moderate NMB, deep neuromuscular blockade improves the surgical space conditions, assessed by the Leiden-Surgical Rating scale, as reported by Martini and colleagues (2).

In this prospective cohort study, we will assess the influence of deep neuromuscular blockade on the surgical space, measured by magnetic resonance imaging (MRI) in patients scheduled for laparoscopic donor nephrectomy

DETAILED DESCRIPTION:
Objective: To establish the influence of deep neuromuscular blockade (NMB) on the abdominal working space during laparoscopy.

Study design: A single center prospective cohort study

Study population: 10 adult patients (18 years or older), equally distributed by gender, scheduled for laparoscopic donor nephrectomy

Study procedures:

Induction of general anesthesia followed by intubation and creation of a pneumoperitoneum (12 mmHg).

Each patient will have a MRI scan during 3 stages:

Phase 1: No neuromuscular blockade (TOF ratio 1) Phase 2: moderate neuromuscular blockade(TOF 1-3). Phase 3: deep neuromuscular blockade (PTC 0-1)

Primary outcome:

The abdominal space measured by MRI: Skin - sacral promontory distance

Secondary outcome:

3D volume measurement of the abdominal cavity by MRI.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for laparoscopic donor nephrectomy
* obtained informed consent

Exclusion Criteria:

* Unable to provide informed consent
* known or suspect allergy to mivacurium, rocuronium or sugammadex
* neuromuscular disease
* indication for rapid sequence induction
* Being unable to undergo MRI due to any reason (e.g. non MRI-compatible implants, epilepsy)
* BMI>30 kg/m2
* American Society of Anesthesiologists (ASA) classification >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Abdominal working space | 3 times (phase 1 (no neuromuscular blockade, phase 2 moderate neuromuscular blockade, phase 3 deep neuromuscular blockade. From start of surgery until third scan, total duration of 30 minutes
  Skin-sacral promontory distance, measured by MRI

SECONDARY OUTCOMES:
Abdominal volume | 3 times (phase 1 no neuromuscular blockade, phase 2 moderate neuromuscular blockade, phase 3 deep neuromuscular blockade. From start of surgery until third scan, total duration of 30 minutes
  3D volume abdominal cavity, measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Michiel C Warlé, Dr., Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bruintjes MH, van Helden EV, Braat AE, Dahan A, Scheffer GJ, van Laarhoven CJ, Warle MC. Deep neuromuscular block to optimize surgical space conditions during laparoscopic surgery: a systematic review and meta-analysis. Br J Anaesth. 2017 Jun 1;118(6):834-842. doi: 10.1093/bja/aex116. PMID 28575335
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Derived] Krijtenburg P, Bruintjes MHD, Futterer JJ, van de Steeg G, d'Ancona F, Scheffer GJ, Keijzer C, Warle MC. MRI measurement of the effects of moderate and deep neuromuscular blockade on the abdominal working space during laparoscopic surgery, a clinical study. BMC Anesthesiol. 2023 Jul 14;23(1):238. doi: 10.1186/s12871-023-02201-1. PMID 37452279